CLINICAL TRIAL: NCT00796614
Title: A Phase IIb/III, Multi-centre, Double-blind, Randomised, Placebo-controlled, Dose Ranging Study of Tamsulosin Hydrochloride (Low, Medium and High Dose) as Treatment in Children With Neuropathic Bladder for Three Months
Brief Title: Study to Evaluate the Efficacy and Safety of Tamsulosin in Children With Neurogenic Bladder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 527.51
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Bladder, Neurogenic
Keywords: tamsulosin; pediatric; neurogenic bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received matching placebo to tamsulosin hydrochloride via opened capsules every day for 14 weeks
  Interventions: Drug: Placebo
- Low dose (Experimental): Participants received 0.001 - 0.002 mg/kg tamsulosin hydrochloride via opened capsules every day for 14 weeks
  Interventions: Drug: tamsulosin hydrochloride
- Medium dose (Experimental): Participants received 0.002 - 0.004 mg/kg tamsulosin hydrochloride via opened capsules every day for 14 weeks
  Interventions: Drug: tamsulosin hydrochloride
- High dose (Experimental): Participants received 0.004 - 0.008 mg/kg tamsulosin hydrochloride via opened capsules every day for 14 weeks
  Interventions: Drug: tamsulosin hydrochloride

INTERVENTIONS:
Drug: tamsulosin hydrochloride — Oral
  Other Names: Flomax; Omnic
  Arms: High dose; Low dose; Medium dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
Aim of this study is to evaluate the efficacy and safety of a range of doses of tamsulosin hydrochloride as treatment in children with an elevated detrusor leak point pressure associated with a known neurological deficit

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic bladder secondary to a known neurologic deficit (e.g. spina bifida)
* Elevated detrusor leak point pressures (LPP) ≥40 cm H2O confirmed by two measurements

Exclusion Criteria:

* Clinically significant abnormalities as determined by the investigator
* A history of relevant orthostatic hypotension, fainting spells or blackouts

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (7):
  - Los Angeles, California
  - Tampa, Florida
  - St Louis, Missouri
  - Buffalo, New York
  - Tarrytown, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
- Ghent, Belgium
- Brazil (2):
  - Santo André
  - São Paulo
- Germany (5):
  - Berlin
  - Deggendorf
  - Essen
  - Hamburg
  - Mainz
- India (13):
  - Ahmedabad
  - Belagavi
  - Bengaluru
  - Hyderabaad
  - Kochi
  - Lucknow
  - Ludhiana
  - Manipal
  - Mumbai
  - Nadiād
  - Nagpur
  - New Delhi
  - Pune
- Italy (3):
  - Cagliari
  - Florence
  - Roma
- Mexico (2):
  - León
  - Puebla City
- Philippines (3):
  - Manila
  - Pasig
  - Quezon City
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Africa (5):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Pretoria
  - Roodepoort
- South Korea (4):
  - Gwangju
  - Incheon
  - Pusan
  - Seoul
- Spain (3):
  - Barcelona
  - Madrid
  - Málaga
- Chernivtsy, Ukraine

REFERENCES:
- See also: Link to Prescribing Information — http://bidocs.boehringer-ingelheim.com/BIWebAccess/ViewServlet.ser?docBase=renetnt&folderPath=/Prescribing+Information/PIs/Flomax+Caps/Flomax.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial included children from 2-16 years of age, with elevated detrusor leak point pressure associated with a known neurologic defect (e.g., spina bifida). The three age strata were 2-<5 years, 5-<10 years and 10-16 years of age. In this study, 231 subjects were enrolled, 162 subjects were randomised and 161 subjects were treated.
Groups:
- Placebo: Subjects were orally administered to matching placebo to tamsulosin hydrochloride, with once daily by sprinkling the content of 2 capsules over a single teaspoonful (5 mL) of apple sauce or yogurt, taken 30 minutes after meal / snack (breakfast). A teaspoonful of water was taken after ingesting the applesauce or yogurt.
- Tamsulosin - Low Dose Level: Subjects were orally administered to low dose level (0.001 - 0.002 mg/kg) of tamsulosin hydrochloride, once daily dependent on a patient's body weight (12.5 kg -100.0 kg), by sprinkling the content of 2 capsules over a single teaspoonful (5 mL) of applesauce or yogurt, taken 30 minutes after meal / snack (breakfast). A teaspoonful of water was taken after ingesting the applesauce or yogurt.
- Tamsulosin - Medium Dose Level: Subjects were orally administered to medium dose level (0.002 - 0.004 mg/kg) of tamsulosin hydrochloride, once daily dependent on a patient's body weight (12.5 kg -100.0 kg), by sprinkling the content of 2 capsules over a single teaspoonful (5 mL) of applesauce or yogurt, taken 30 minutes after meal / snack (breakfast). A teaspoonful of water was taken after ingesting the applesauce or yogurt.
- Tamsulosin - High Dose Level: Subjects were orally administered to high dose level (0.004 - 0.008 mg/kg) of tamsulosin hydrochloride, once daily dependent on a patient's body weight (12.5 kg -100.0 kg), by sprinkling the content of 2 capsules over a single teaspoonful (5 mL) of applesauce or yogurt, taken 30 minutes after meal / snack (breakfast). A teaspoonful of water was taken after ingesting the applesauce or yogurt.
Period: Overall Study
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Started | 41 | 40 | 39 | 41
Not Treated | 0 | 0 | 1 | 0
Completed | 36 | 36 | 36 | 40
Not Completed | 5 | 4 | 3 | 1
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Other than stated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Includes all patients who were documented to have taken at least one dose of randomised treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level | Total
Number analyzed (Participants) | 41 | 40 | 39 | 41 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.4 (3.7) | 8.1 (4.2) | 8.1 (3.8) | 8.2 (4.3) | 8.2 (4.0)
Age, Customized [Number; unit: participants]
  2 to < 5 years | 7 | 8 | 7 | 8 | 30
  5 to < 10 years | 18 | 17 | 17 | 18 | 70
  10 to 16 years | 16 | 15 | 15 | 15 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 14 | 16 | 64
  Male | 25 | 22 | 25 | 25 | 97

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment Defined as Patients Who Decrease Their Detrusor Leak Point Pressure (LPP) to <40 cm H2O Based Upon Two Evaluations on the Same Day.
Description: The primary endpoint was response to treatment defined as patients who decreased their detrusor leak point pressure (LPP) based upon two evaluations on the same day to less than 40 cm H2O at Week 14 (end of treatment). Detrusor leak point pressure (LPP) recorded in cm H2O was obtained using a standard urodynamic technique, a cystometrogram. On treatment (OT): Consist of all on treatment data. Observations measured ≤3 days of stopping treatment was considered as on treatment. Missing data in these analyses was not replaced or imputed.
Time Frame: Week 14
Population: Full analysis set-LPP (FAS-LPP): Includes all patients in the treated set who received at least one dose of randomised. FAS-LPP contains same patients as TS.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 34 | 35 | 33 | 33
Percentage of participants | 35.3 | 45.7 | 27.3 | 42.4
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; Logistic regression model was used with treatment variable and three covariates: age group, concomitant use of anti-cholinergic medication and geographic region. The first two covariates were used in the stratification of the randomisation. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.5388, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.50 to 3.80]
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3430, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.20 to 1.76]
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5209, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.50 to 3.97]
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin - Low Dose Level vs Tamsulosin - Medium Dose Level vs Tamsulosin - High Dose Level; A test of trend across the four treatment groups was performed as a secondary analysis in the proportion of responders across the dose levels using Cochran-Armitage trend test; Test type: Superiority or Other; p = 0.9436, Cochran-Armitage trend test

2. Secondary Outcome: Change From Baseline in LPP at Week 14 (End of Treatment)
Description: Change from baseline in detrusor leak point pressure (LPP) at Week 14 (end of treatment) between each dose group and the placebo group was compared for the FAS-LPP.
Time Frame: Baseline and Week 14
Population: Full analysis set-LPP (FAS-LPP), OT
Measure: Least Squares Mean (Standard Error); unit: cm H2O
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 30 | 32 | 31 | 33
cm H2O | -11.4 (4.6) | -17.6 (4.5) | -4.6 (4.4) | -14.3 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; ANCOVA model was used with covariates of age group, anti-cholinergic use at baseline and geographic region. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.3097, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2676, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6265, ANCOVA

3. Secondary Outcome: Percentage Change From Baseline in LPP at Week 14 (End of Treatment)
Description: Percent changes in detrusor leak point pressure (LPP) from baseline to the end of treatment at Week 14 between each dose group and the placebo group were compared for the FAS-LPP.
Time Frame: Baseline and Week 14.
Population: Full analysis set-LPP (FAS-LPP), OT
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 30 | 32 | 31 | 33
Percentage change | -19.9 (7.3) | -27.4 (7.1) | -1.9 (7) | -23.9 (6.9)
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4359, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0658, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6709, ANCOVA

4. Secondary Outcome: Response With Regard to Hydronephrosis Was Defined as Improvement or Stabilisation Based Upon the Renal Ultrasound Grading at Week 14 (End of Treatment) Compared to Baseline
Description: Hydronephrosis response was defined as stabilisation or improvement of hydronephrosis measured by renal ultrasound at the end of treatment when compared to baseline, based on ultrasound grading.
  The lower or same grade at end of treatment compared to baseline is considered an improvement or stabilization
Time Frame: Baseline and Week 14
Population: Full analysis set-renal (FAS-RENAL): This analysis set includes all patients in the treated set who received at least one dose of randomised treatment and had at least one on-treatment renal ultrasound measurement.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 40 | 38 | 38 | 40
Participants
  Left Kidney [N= 34; 34; 33; 40] | 32 | 31 | 31 | 37
  Right Kidney [N= 33; 34; 34; 40] | 31 | 33 | 30 | 38
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; Patient responded to tamsulosin-low dose (Left Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.5672, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; Patient responded to tamsulosin-medium dose (Left Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.8724, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; Patient responded to tamsulosin-high dose (Left Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.7674, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin - Low Dose Level; Patient responded to tamsulosin-low dose (Right Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.5545, Regression, Logistic
Statistical Analysis 5: Comparison: Placebo vs Tamsulosin - Medium Dose Level; Patient responded to tamsulosin-Medium dose (Right Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.4774, Regression, Logistic
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin - High Dose Level; Patient responded to tamsulosin-High dose (Right Kidney) was compared to placebo. Logistic regression model was used with age group, anti-cholinergic use,and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.8626, Regression, Logistic

5. Secondary Outcome: Response With Regard to Hydroureter Was Defined as Improvement or Stabilisation Based Upon the Renal Ultrasound at Week 14 (End of Treatment) Compared to Baseline
Description: Hydroureter response was defined as stabilisation or improvement based on change from baseline in the presence or absence of hydroureter at the end of treatment (Week 14).
  Response defined as stabilization or improvement of hydroureter measured by renal ultrasound compared to baseline by treatment group (Patients are classified according to the treatment they were taking at Week 14 or end of treatment) at Week 14.
Time Frame: Baseline and Week 14
Population: Full analysis set-renal (FAS-RENAL)
Measure: Number; unit: Participants
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 40 | 38 | 38 | 40
Participants
  Left Kidney (N= 34, 34, 33, 40) | 33 | 33 | 32 | 38
  Right Kidney (N= 33, 34, 34, 40) | 33 | 33 | 32 | 38
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9669, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.9231, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.6360, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs Tamsulosin - Low Dose Level; Patient responded to tamsulosin-low dose (Right Kidney) was compared to placebo. Fisher's exact test was used for this analysis; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 5: Comparison: Placebo vs Tamsulosin - Medium Dose Level; Patient responded to tamsulosin-medium dose (Right Kidney) was compared to placebo. Fisher's exact test was used for this analysis; Test type: Superiority or Other; p = 0.4925, Fisher Exact
Statistical Analysis 6: Comparison: Placebo vs Tamsulosin - High Dose Level; Patient responded to tamsulosin-high dose (Right Kidney) was compared to placebo. Fisher's exact test was used for this analysis; Test type: Superiority or Other; p = 0.4977, Fisher Exact

6. Secondary Outcome: Change From Baseline in Urine Volume at Week 14
Description: Change in baseline urine volumes obtained by catheterisation as recorded in catheterisation diary at Week 14.
Time Frame: Baseline and Week 14
Population: Full analysis set-catheter (FAS-CATH): This analysis set includes all patients in the treated set who received at least one dose of randomised treatment, were on a catheterisation regimen, and had at least one on-treatment catheterisation assessment.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 24 | 18 | 16 | 21
mL | -2.3 (14.0) | -32.2 (15.5) | 4.4 (16.3) | 3.3 (14.2)
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; ANCOVA model was used with age group, anti-cholinergic use, and geographic region as covariates. On treatment (OT) analyses approach was used; Test type: Superiority or Other; p = 0.1373, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.7440, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.7703, ANCOVA

7. Secondary Outcome: Change From Baseline in Number of Times Patient Was Wet at Catheterisation
Description: Change from baseline in number of times patient was wet at time of catheterisation as recorded in catheterisation diary.
Time Frame: Baseline and Week 14
Population: Full analysis set-catheter (FAS-CATH)
Measure: Least Squares Mean (Standard Error); unit: Times patient wet at catheterization
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 24 | 18 | 16 | 21
Times patient wet at catheterization | 0.3 (0.8) | -1.7 (0.9) | 0.0 (0.9) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Tamsulosin - Low Dose Level; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0808, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Tamsulosin - Medium Dose Level; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.8244, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Tamsulosin - High Dose Level; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.5045, ANCOVA

8. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic Testing, Electorocardiogram (ECG), Laboratory Values, Urinalysis, Treatment Emergent AE's and Cognitive Testing.
Description: Number of participants with Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic testing (blood pressure, pulse and respiratory rate), Electrocardiogram (ECG), Laboratory Values inclusive of hormonal assays, vision testing, Cognitive Testing, Occurrence of treatment emergent adverse events, Premature discontinuation of study drug due to AE and Urinalysis.
  Relevant findings or worsening of baseline conditions were reported as adverse events.
Time Frame: From first drug administration until 28 days after last study drug administration, upto 160 days
Population: Treated Set (TS).
  All subjects began treatment with their low dose and then they were titrated to their randomised medium or high dose. Therefore some of the subjects were counted more than once for having reported adverse events with different doses of the study.
Measure: Number; unit: Participants
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 41 | 120 | 80 | 40
Participants
  Occurrence of treatment emergent adverse events | 18 | 39 | 24 | 15
  Premature discontinuation of study drug due to AE | 1 | 2 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 1

9. Secondary Outcome: Post Void Residual Volume at Week 14
Description: Median change from baseline to Week 14 in post void residual (mL) by study treatment.
Time Frame: Baseline and Week 14.
Population: Treated Set (TS). Number of particiapants Analysed are the number of participants whose data were available for this endpoint.
Measure: Median (Standard Deviation); unit: mL
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Number analyzed (Participants) | 31 | 36 | 34 | 38
mL | 3 (80.28) | -19 (66.4) | -1.5 (92.33) | 0.00 (58.67)

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last study drug administration, upto 160 days.
Description: All subjects began treatment with their low dose and then they were titrated to their randomised medium or high dose. Therefore some of the subjects were counted more than once for having reported adverse events with different doses of the study.
Arm/Group | Placebo | Tamsulosin - Low Dose Level | Tamsulosin - Medium Dose Level | Tamsulosin - High Dose Level
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/120 | 0/80 | 0/40
Other Adverse Events (participants affected / at risk) | 13/41 | 19/120 | 14/80 | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Tamsulosin - Low Dose Level (N=120) | Tamsulosin - Medium Dose Level (N=80) | Tamsulosin - High Dose Level (N=40)
Death (General disorders) | 0 | 1 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Tamsulosin - Low Dose Level (N=120) | Tamsulosin - Medium Dose Level (N=80) | Tamsulosin - High Dose Level (N=40)
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 4 | 3
Influenza (Infections and infestations) | 3 | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 5 | 4 | 4
Urinary tract infection (Infections and infestations) | 4 | 8 | 2 | 5
Headache (Nervous system disorders) | 6 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 0

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.